CLINICAL TRIAL: NCT04699461
Title: A Phase 2 Randomized Study of Loncastuximab Tesirine Versus Idelalisib in Patients With Relapsed or Refractory Follicular Lymphoma (LOTIS-6)
Brief Title: Study to Evaluate the Efficacy and Safety of Loncastuximab Tesirine Versus Idelalisib in Participants With Relapsed or Refractory Follicular Lymphoma
Acronym: LOTIS-6
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative decision (not due to safety reason)
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADCT 402-202; 2020-003695-40 (EudraCT Number)
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Relapsed Follicular Lymphoma; Refractory Follicular Lymphoma
Keywords: Relapsed Follicular Lymphoma; Refractory Follicular Lymphoma; Loncastuximab Tesirine; Follicular Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — loncastuximab tesirine; idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Loncastuximab Tesirine (Experimental): Participants will be administered loncastuximab tesirine as an intravenous (IV) infusion on Day 1 of each cycle, where 1 cycle is 3 weeks. Loncastuximab tesirine will be administered at a dose of 150 μg/kg for 2 cycles, then at a dose of 75 μg/kg for subsequent cycles.
  Interventions: Drug: Loncastuximab Tesirine
- Idelalisib (Active Comparator): Participants will be administered 150 mg idelalisib, orally, twice a day throughout each cycle, where 1 cycle is 4 weeks.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Loncastuximab Tesirine — IV infusion
  Other Names: Zynlonta; ADCT-402
  Arms: Loncastuximab Tesirine
Drug: Idelalisib — Oral tablet
  Arms: Idelalisib

SUMMARY:
This study aims to evaluate the efficacy of single agent loncastuximab tesirine compared to idelalisib in participants with relapsed or refractory follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any study procedures.
* Male or female participants aged 18 years or older, with pathologic diagnosis of follicular lymphoma (FL) (Grade 1, 2, 3A) in the most recent tumor biopsy.
* Relapsed or refractory disease following two or more treatment regimens, at least one of which must have contained an anti-CD20 therapy.
* Participants who have received previous CD19-directed therapy must have a biopsy which shows CD19 expression after completion of the CD19-directed therapy.
* Measurable disease as defined by the 2014 Lugano Classification as assessed by positron emission tomography - computed tomography (PET-CT) or, if not Fluorodeoxyglucose (FDG) avid, CT or magnetic resonance imaging (MRI).
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block (or minimum 10 freshly cut unstained slides if block is not available). Note: Any biopsy since initial diagnosis is acceptable, but if several samples are available, the most recent sample is preferred.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Adequate organ function as defined by screening laboratory values within the following parameters:

  1. Absolute neutrophil count (ANC) ≥1.0 × 10^3/μL (off growth factors at least 72 hours),
  2. Platelet count ≥75 × 10^3/μL without transfusion in the past 2 weeks,
  3. Alanine aminotransferase, AST, and GGT ≤2.5 × the upper limit of normal (ULN),
  4. Total bilirubin ≤1.5 × ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 × ULN),
  5. Calculated creatinine clearance ≥30 mL/min by the Cockcroft and Gault equation. Note: A laboratory assessment may be repeated a maximum of two times during the Screening period to confirm eligibility
* Women of childbearing potential (WOCBP)(1) must agree to use a highly effective method(2) of contraception from the time of giving informed consent until at least 9 months after the last dose of study treatment. Men with female partners who are of childbearing potential must agree to use a condom when sexually active or practice total abstinence from the time of giving informed consent until at least 6 months after the participant receives his last dose of study treatment.

  1. WOCBP are defined as sexually mature women who have not undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or who have not been postmenopausal. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
  2. Highly effective forms of birth control are methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Highly effective forms of birth control include hormonal contraceptives associated with inhibition of ovulation (oral, injectable, patch, intrauterine devices), male partner sterilization, or total abstinence from heterosexual intercourse, when this is the preferred and usual lifestyle of the participant.

Note: The double-barrier method (e.g., synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), periodic abstinence (such as calendar, symptothermal, post ovulation), withdrawal (coitus interruptus), lactational amenorrhea method, and spermicide-only are not acceptable as highly effective methods of contraception.

Exclusion Criteria:

* Previous treatment with loncastuximab tesirine.
* Previous treatment with idelalisib.
* History of hypersensitivity to any of the excipients of loncastuximab tesirine or idelalisib.
* Follicular lymphoma which has transformed to diffuse large B-cell lymphoma (DLBCL) or other aggressive lymphomas.
* Requires treatment or prophylaxis with a strong cytochrome P450 (CYP) 3A inhibitor, inducer, or sensitive substrate.
* History of or ongoing drug-induced pneumonitis.
* History of or ongoing inflammatory bowel disease.
* Any condition that could interfere with the absorption or metabolism of idelalisib including malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
* Active second primary malignancy other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary.
* Autologous transplant within 30 days prior to start of study treatment (C1D1).
* Allogenic transplant within 60 days prior to start of study treatment (C1D1).
* Active graft-versus-host disease.
* Post-transplantation lymphoproliferative disorders.
* Human immunodeficiency virus (HIV) seropositive with any of the following:

  1. CD4+ T-cell counts <350 cells/μL.
  2. Acquired immuno-deficiency syndrome (AIDS)-defining opportunistic infection within 12 months prior to screening.
  3. Not on anti-retroviral therapy, or on anti-retroviral therapy for < 4 weeks at the time of screening.
  4. HIV viral load ≥400 copies/mL.
* Serologic evidence of chronic hepatitis B infection and unable or unwilling to receive standard prophylactic anti-viral therapy or with detectable hepatitis B virus (HBV) viral load.
* Serologic evidence of hepatitis C infection without completion of curative treatment or with detectable hepatitis C virus (HCV) viral load.
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
* Lymphoma with active central nervous system involvement, including leptomeningeal disease.
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
* Breastfeeding or pregnant.
* Significant medical comorbidities, including but not limited to, uncontrolled hypertension (BP ≥160/100 mm Hg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes, or severe chronic pulmonary disease.
* Any Grade ≥3 active infection which requires IV antibiotics, IV antiviral, or IV antifungal treatment.
* Major surgery, radiotherapy, chemotherapy or other anti-neoplastic therapy within 14 days prior to start of study treatment (C1D1), except shorter if approved by the Sponsor.
* Use of any other experimental medication within 30 days prior to start of study treatment (C1D1).
* Live vaccine administration within 4 weeks prior to Cycle(C) 1 Day (D) 1.
* Failure to recover to ≤ Grade 1 (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) from acute non-hematologic toxicity (except ≤Grade 2 neuropathy or alopecia) due to previous therapy prior to screening.
* Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the participant inappropriate for study participation or put the participant at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (5):
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group - Florham Park Campus, Florham Park, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Hollings Cancer Center, Charleston, South Carolina
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire Universite Catholique de Louvain, Yvoir
- France (4):
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier de La Rochelle, La Rochelle
  - Centre de Lutte Contre le Cancer - Centre Henri-Becquerel, Rouen
  - Hôpital Bretonneau, Tours
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Pécsi Tudományegyetem Klinikai Központ, Pécs
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Carmel Medical Center, Haifa
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Azienda Ospedaliero - Universitaria Careggi, Florence, Italy
- Poland (3):
  - Szpitale Pomorskie Spółka Z Ograniczoną Odpowiedzialnością, Gdynia
  - Pratia Onkologia Katowice, Katowice
  - Pratia Poznań, Skorzewo
- Spain (8):
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), L'Hospitalet de Llobregat
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Virgen del Rocío, Seville
- Inselspital Universitätsspital Bern, Bern, Switzerland
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Account University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Loncastuximab Tesirine: Participants were administered loncastuximab tesirine as an intravenous (IV) infusion on Day 1 of each cycle, where 1 cycle is 3 weeks. Loncastuximab tesirine will be administered at a dose of 150 μg/kg for 2 cycles, then at a dose of 75 μg/kg for subsequent cycles.
  The median number of treatment cycles was 5.5 (min: 5; max: 12). The median treatment duration was 122.5 days (min: 54; max: 231 days).
- Idelalisib: Participants were administered 150 mg idelalisib, orally, twice a day throughout each cycle, where 1 cycle is 4 weeks.
  1 participant received 6 cycles and the other participant received 13 cycles of treatment. The treatment duration was 140 days and 333 days, respectively.
Period: Overall Study
Arm/Group | Loncastuximab Tesirine | Idelalisib
Started | 4 | 2
Completed | 0 | 0
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study termination by sponsor | 2 | 1
Not completed — Death | 1 | 0
Not completed — Radiographic progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Loncastuximab Tesirine: Participants were administered loncastuximab tesirine as an intravenous (IV) infusion on Day 1 of each cycle, where 1 cycle is 3 weeks. Loncastuximab tesirine was administered at a dose of 150 μg/kg for 2 cycles, then at a dose of 75 μg/kg for subsequent cycles.
  The median number of treatment cycles was 5.5 (min: 5; max: 12). The median treatment duration was 122.5 days (min: 54; max: 231 days).
- Total: Total of all reporting groups
Arm/Group | Loncastuximab Tesirine | Idelalisib | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Customized [Count of Participants; unit: Participants]
  55 to 69 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR)
Description: CRR was defined as the percentage of participants who experienced a best overall response (BOR) of complete response (CR) assessed prior to any subsequent anticancer treatment.
Time Frame: Up to the end of treatment, maximum time on treatment was 333 days
Population: No response data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a BOR of CR or partial response (PR) assessed prior to any subsequent anticancer treatment.
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No response data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time between the randomization date and the first documentation of recurrence, progression, or death.
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: Inclusive of participants who experienced recurrence, progression, or death.
Measure: Median (Full Range); unit: days
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 1 | 1
days | NA [NA to NA] — Due to risk of re-identification. | NA [NA to NA] — Due to risk of re-identification.

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the randomization date and death from any cause.
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: Inclusive of participants who experienced death.
Measure: Median (Full Range); unit: days
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 1 | 0
days | NA [NA to NA] — Due to risk of re-identification. |

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the documentation of tumor response to disease progression or death.
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No response data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Event (TEAE)
Description: TEAEs were defined as an AE that occurs or worsens in the period extending from the first dose of study treatment until 30 days after the last dose of study treatment or start of new anti-cancer therapy, whichever is earlier.
  Any clinically significant changes from baseline in the safety laboratory values, vital signs, 12-lead electrocardiogram (ECG), and Eastern Cooperative Oncology Group (ECOG) performance status were reported as TEAEs.
Time Frame: Day 1 to 30 days after end of treatment, maximum time on treatment was 333 days
Measure: Count of Participants; unit: Participants
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 4 | 2
Participants
  TEAEs | 4 | 2
  Serious TEAEs | 3 | 0

7. Secondary Outcome: Average Concentration of Loncastuximab Tesirine Before Infusion
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Average Concentration of Loncastuximab Tesirine at the End of Infusion
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Clearance Rate of Loncastuximab Tesirine
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Volume of Distribution of Loncastuximab Tesirine
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Titers to Loncastuximab Tesirine
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Measured by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L)
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Measured by the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym)
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Specific Symptomatic Adverse Event Symptoms As Selected From Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The specific symptomatic adverse events includes fatigue, swelling, rash, nausea, diarrhea, abdominal pain, and cough.
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Treatment-Related Symptoms as Assessed by Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The specific symptoms assessed include fatigue, swelling, rash, nausea, diarrhea, abdominal pain, and cough. The severity is assessed from "None" to "Very severe" and the interference level is assessed from "Not at all" to "Very much."
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Population: No data was collected.
Arm/Group | Loncastuximab Tesirine | Idelalisib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to end of treatment, maximum time on treatment was 333 days
Arm/Group | Loncastuximab Tesirine | Idelalisib
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/4 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Loncastuximab Tesirine (N=4) | Idelalisib (N=2)
Anemia (Blood and lymphatic system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Loncastuximab Tesirine (N=4) | Idelalisib (N=2)
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 0
COVID-19 infection (Infections and infestations) | 2 | 1
Asthenia (General disorders) | 1 | 0
Blood creatinine increased, (Investigations) | 0 | 1
Dysphagia, (General disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Porphyria non-acute (Hepatobiliary disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Neutropenia (Investigations) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was terminated (administrative decision) by the sponsor following the withdrawal of idelalisib from the US market for the relapsed FL indication (i.e., not due to any safety reasons emerging from this study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04699461/Prot_SAP_000.pdf